CLINICAL TRIAL: NCT03174743
Title: The Effect of Protective Ventilation During Pulmonary Lobectomy
Brief Title: Protective Ventilation During Pulmonary Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Su Liu, Principal Investigator, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYFY-2017-033
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Complication; Thoracic Surgery; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Convential Ventilation 1 (Placebo Comparator): Intraoperatively ventilated patients with a tidal volume (VT) of 10 ml/kg of ideal body weight, the level of PEEP at 0 cmH2O and a FiO2 of 60%.
  Interventions: Procedure: Convential Ventilation 1
- Convential Ventilation 2 (Placebo Comparator): Intraoperatively ventilated patients with a tidal volume (VT) of 10 ml/kg of ideal body weight, the level of PEEP at 0 cmH2O and a FiO2 of100%.
  Interventions: Procedure: Convential Ventilation 2
- Protective ventilation 1 (Active Comparator): Intraoperatively ventilated patients with a tidal volume (VT) of 6 ml/kg of ideal body weight, the level of PEEP at 6 cmH2O and a FiO2 of 60% with lung recruitment maneuvers.
  Interventions: Procedure: Protective Ventilation 1
- Protective ventilation 2 (Active Comparator): Intraoperatively ventilated patients with a tidal volume (VT) of 6 ml/kg of ideal body weight, the level of PEEP at 6 cmH2O and a FiO2 of 100% with lung recruitment maneuvers.
  Interventions: Procedure: Protective Ventilation 2

INTERVENTIONS:
Procedure: Convential Ventilation 1 — High tidal volume, moderate inspired oygen fraction (FiO2).
  Arms: Convential Ventilation 1
Procedure: Convential Ventilation 2 — High tidal volume, high inspired oygen fraction (FiO2).
  Arms: Convential Ventilation 2
Procedure: Protective Ventilation 1 — Low tidal volume, PEEP, moderate inspired oygen fraction (FiO2) and recruitment maneuver.
  Arms: Protective ventilation 1
Procedure: Protective Ventilation 2 — Low tidal volume, PEEP, High inspired oygen fraction (FiO2) and recruitment maneuver.
  Arms: Protective ventilation 2

SUMMARY:
The investigator will evaluate the influence of lung protective ventilation on postoperative clinical outcome in patients undergoing one-lung ventilation for pulmonary lobectomy.

DETAILED DESCRIPTION:
The hypothesis is that application of low tidal volume, moderate inspired oxygen fraction (FiO2) ,intermittent alveolar recruitment and positive end-expiratory pressure (PEEP) would be more beneficial than conventional ventilation in patients.

ELIGIBILITY:
Inclusion Criteria:

1.20 Years and older 2.Patients undergoing pulmonary lobectomy

Exclusion Criteria:

1. Emergency surgery
2. Pulmonary hypertension
3. Forced vital capacity or forced expiratory volume in 1 sec < 50% of the predicted values
4. Coagulation disorder
5. Pulmonary or extrapulmonary infections
6. History of treatment with steroid in 3 months before surgery
7. History of recurrent pneumothorax
8. History of lung resection surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with pulmonary complication | up to postoperative 3days
  The number of patients with pulmonary complication including atelectasis, pulmonary infiltration, pulmonary edema, pulmonary infection, pleural effusion and pulmonary embolism.

SECONDARY OUTCOMES:
PaO2 /FiO2 | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation, 1 hour after the end of surgery
respiratory compliance | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  Dynamic compliance, Static compliance
IL6 | 10 min after induction, 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
IL10 | 10 min after induction, 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Liu Su Liu, M.D/Ph.D, Principal Investigator — 徐州医科大学附属医院医学
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published.

REFERENCES:
- [Result] Theroux MC, Fisher AO, Horner LM, Rodriguez ME, Costarino AT, Miller TL, Shaffer TH. Protective ventilation to reduce inflammatory injury from one lung ventilation in a piglet model. Paediatr Anaesth. 2010 Apr;20(4):356-64. doi: 10.1111/j.1460-9592.2009.03195.x. Epub 2009 Nov 16. PMID 19919624
- [Result] Fuller BM, Mohr NM, Drewry AM, Carpenter CR. Lower tidal volume at initiation of mechanical ventilation may reduce progression to acute respiratory distress syndrome: a systematic review. Crit Care. 2013 Jan 18;17(1):R11. doi: 10.1186/cc11936. PMID 23331507
- [Result] Kozian A, Schilling T, Schutze H, Senturk M, Hachenberg T, Hedenstierna G. Ventilatory protective strategies during thoracic surgery: effects of alveolar recruitment maneuver and low-tidal volume ventilation on lung density distribution. Anesthesiology. 2011 May;114(5):1025-35. doi: 10.1097/ALN.0b013e3182164356. PMID 21436678
- [Result] Licker M, Diaper J, Villiger Y, Spiliopoulos A, Licker V, Robert J, Tschopp JM. Impact of intraoperative lung-protective interventions in patients undergoing lung cancer surgery. Crit Care. 2009;13(2):R41. doi: 10.1186/cc7762. Epub 2009 Mar 24. PMID 19317902
- [Result] Ishikawa S. Alveolar recruitment maneuver as an important part of protective one-lung ventilation. J Anesth. 2012 Oct;26(5):794-5. doi: 10.1007/s00540-012-1396-4. Epub 2012 May 3. No abstract available. PMID 22552387
- [Result] Yang M, Ahn HJ, Kim K, Kim JA, Yi CA, Kim MJ, Kim HJ. Does a protective ventilation strategy reduce the risk of pulmonary complications after lung cancer surgery?: a randomized controlled trial. Chest. 2011 Mar;139(3):530-537. doi: 10.1378/chest.09-2293. Epub 2010 Sep 9. PMID 20829341
- [Result] Kim SH, Jung KT, An TH. Effects of tidal volume and PEEP on arterial blood gases and pulmonary mechanics during one-lung ventilation. J Anesth. 2012 Aug;26(4):568-73. doi: 10.1007/s00540-012-1348-z. Epub 2012 Feb 18. PMID 22349751
- [Result] Ahn HJ, Kim JA, Yang M, Shim WS, Park KJ, Lee JJ. Comparison between conventional and protective one-lung ventilation for ventilator-assisted thoracic surgery. Anaesth Intensive Care. 2012 Sep;40(5):780-8. doi: 10.1177/0310057X1204000505. PMID 22934859